CLINICAL TRIAL: NCT05065138
Title: Comparison of the Effect of Helicobacter Pylori Eradication Before and After the Training of Gastroenterologists on Standardized Helicobacter Pylori Eradication Therapy
Brief Title: Comparison of Helicobacter Pylori Eradication Effect Before and After Training of Gastroenterologists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, doctoral supervisor of Qilu Hospital gastroenterology department, Shandong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021SDU-QILU-G004-2
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Standardized training on Helicobacter pylori eradication; Gastroenterologist

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- After receiving standardized training on Helicobacter pylori eradication (Experimental): After the gastroenterologists receive standardized training to eradicate Helicobacter pylori, they recruit Helicobacter pylori-positive patients for treatment.
  Interventions: Behavioral: Standardized training on Helicobacter pylori eradication treatment
- Before receiving standardized training on Helicobacter pylori eradication (No Intervention): Gastroenterologists recruited patients with Helicobacter pylori positive for treatment before receiving standardized training on Helicobacter pylori eradication.

INTERVENTIONS:
Behavioral: Standardized training on Helicobacter pylori eradication treatment — Standardized training on Helicobacter pylori eradication treatment
  Arms: After receiving standardized training on Helicobacter pylori eradication

SUMMARY:
The researchers recruited gastroenterologists. Physician subjects recruited Helicobacter pylori-positive patients before and after receiving standardized training on Helicobacter pylori eradication. There are no restrictions on treatment options and drugs during the trial. Compare the eradication rate, adverse reaction rate, and patient compliance before and after physician training.

DETAILED DESCRIPTION:
The researchers recruited no less than 20 gastroenterologists to participate in the study, and gastroenterologists recruited 25 patients who were over 18 years of age and were positive for Helicobacter pylori for the first time. In this process, the patient population is not restricted, and the eradication program is not restricted. Gastroenterologists followed up their diagnosis and treatment. Researchers track and record patients' medications and adverse reactions during medication via phone or WeChat to assess patient compliance. Record the eradication rate. The researchers will provide standardized Helicobacter pylori eradication training for the Department of Gastroenterology after all patients treated by gastroenterologists have been eradicated and reviewed. After the training, the gastroenterologist recruited 25 patients who were over 18 years old and were newly treated with Helicobacter pylori positive. In this process, the patient population is not restricted, and the eradication program is not restricted. Gastroenterologists followed up their diagnosis and treatment. Researchers track and record patients' medications and adverse reactions during medication via phone or WeChat to assess patient compliance. Record the eradication rate. Compare the eradication rate, adverse reaction rate and compliance of patients before and after the training of gastroenterologists.

ELIGIBILITY:
Inclusion Criteria:

* 1.Physician specialized in gastroenterology.
* 2.Diagnosis and treatment conditions for H. pylori exist in the hospital where the gastroenterology doctor is located.

(C13 urea breath test, C14 urea breath test, rapid urease test, stool H. pylori antigen test, histopathological test, H. pylori culture, any of the above)

Exclusion Criteria:

* 1.Those who are unable or unwilling to provide informed consent.
* 2.Patients with H. pylori have never been diagnosed and treated.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1025 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Eradication rate | 1 year
  The eradication rate of before and after the gastroenterologists receiving

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Xiuli Zuo, Jinan, Shandong, China